CLINICAL TRIAL: NCT00053040
Title: Phase I/II Trial Of Intracerebral IL13-PE38QQR Infusions In Pediatric Patients With Recurrent Malignant Glioma
Brief Title: Immunotoxin Therapy in Treating Children With Recurrent Malignant Gliomas
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Withdrawal of pharmaceutical company support for the investigational drug
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: James M. Boyett/PBTC Operations and Biostatistics Center Executive Director, Pediatric Brain Tumor Consortium
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000269073; PBTC-011C (Other: Pediatric Brain Tumor Consortium); NEOPHARM-IL13PEI-151 (Other: Neopharm); NCI-5930 (Other: NCI)
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent childhood brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — IL13-PE38

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Surgery for tumor resection + IL13-PE38QQR infusion (Experimental)
  Interventions: Biological: cintredekin besudotox; Procedure: conventional surgery

INTERVENTIONS:
Biological: cintredekin besudotox — IL13-PE38QQR is administered intracerebrally by continuous convection enhanced infusion at a starting concentration of 0.25 μg/mL. Infusion duration will be held constant at 96 hours (4 days). The phase I component of this study is to estimate the maximum safe total flow rate and the maximum safe infusion concentration.
  Other Names: IL13-PE38QQR
Procedure: conventional surgery — Conventional surgery is used for tumor resection prior to catheter placement for IL13-PE38QQR infusion.

SUMMARY:
RATIONALE: Immunotoxins can locate tumor cells and kill them without harming normal cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of immunotoxin therapy and to see how well it works in treating children undergoing surgery for recurrent or progressive malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the toxicity of peritumoral IL13-PE38QQR after surgical resection in pediatric patients with recurrent malignant gliomas. (Phase I)
* Determine the maximum tolerated flow rate and maximum tolerated infusion concentration (MTiC) of this drug in these patients. (Phase I)
* Estimate the rate of survival after initial progression in patients treated at the maximum safe flow rate and MTiC with this drug. (Phase II)

Secondary

* Describe the overall safety and tolerability of this regimen in these patients from the start of infusion through disease progression or initiation of alternative treatment.
* Determine the IL13 receptor α2 chain expression status and distribution in pediatric recurrent or progressive malignant gliomas
* Estimate the progression-free survival of patients treated with this drug. (Phase II)

OUTLINE: This is a multicenter, dose-escalation study.

* Phase I: Patients undergo surgical resection of the tumor. Within 2-7 days later, patients undergo placement of 2-4 peritumoral catheters. One to 2 days later, patients receive peritumoral IL13-PE38QQR continuously over 96 hours. Catheters are removed after completion of the infusion.

Cohorts of 3 patients receive IL13-PE38QQR at escalating flow rates and a fixed concentration until the maximum safe flow rate is determined. The maximum safe flow rate is defined as the rate prior to the one at which 2 of 3 or more patients experience dose-limiting toxicity.

Following determination of the maximum safe flow rate, cohorts of 2-3 patients receive IL13-PE38QQR at escalating concentrations at the maximum safe flow rate until the maximum tolerated infusion concentration (MTiC) is determined. The MTiC is defined as the concentration prior to the one at which 2 of 3 or more patients experience dose-limiting toxicity.

* Phase II: Patients receive IL13-PE38QQR as above at the maximum safe flow rate and MTiC determined in the phase I of the study.

Patients are followed at week 18 after catheter placement and then every 8 weeks thereafter until death, disease progression, or completion of six months (phase I) or 12 months (phase II) of follow-up after the end of IL13-PE38QQR infusion. Phase II patients who complete one year of follow-up without disease progression are followed every 12 weeks thereafter until death.

PROJECTED ACCRUAL: Approximately 2-50 patients (2-24 for phase I and approximately 26 for phase II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed grade 3 or 4 supratentorial malignant glioma by prior surgery or biopsy

  * Anaplastic astrocytoma
  * Glioblastoma multiforme
  * Malignant mixed oligoastrocytoma
* Recurrent or progressive disease by radiology

  * In first progression or recurrence (for patients in the phase II portion of the study only)
* Must have 1 solid primary lesion with a solid component measuring at least 1 cm in diameter
* Must have received external beam radiotherapy with tumor dose of at least 48 Gy
* Planning to undergo gross total resection of the tumor to remove all contrast-enhancing components of the tumor

  * No multifocal tumor not amenable to gross tumor resection
* No contrast-enhancing tumor component crossing the midline
* No subependymal or leptomeningeal tumor dissemination
* No clinically significant increased intracranial pressure (e.g., impending herniation)
* No spinal cord compression
* No requirement for immediate palliative treatment

PATIENT CHARACTERISTICS:

Age

* 3 to 21

Performance status

* Karnofsky 60-100% (over 16 years of age)
* Lansky 60-100 (16 years of age and under)

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Hemoglobin at least 10 g/dL*
* Platelet count at least 100,000/mm^3* NOTE: *Transfusion independent

Hepatic

* PT and PTT normal

Renal

* Creatinine normal for age

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled seizures

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 8 weeks since prior hematopoietic stem cell transplantation

Chemotherapy

* No prior intracerebral chemotherapy for malignant glioma (except polifeprosan 20 with carmustine implant)
* At least 6 months since prior polifeprosan 20 with carmustine implant
* At least 4 weeks since prior cytotoxic chemotherapy (6 weeks for nitrosoureas)
* At least 2 weeks since prior vincristine or noncytotoxic chemotherapy
* No concurrent chemotherapy

Endocrine therapy

* Concurrent steroids allowed

Radiotherapy

* See Disease Characteristics
* At least 8 weeks since prior radiotherapy
* No prior focal radiotherapy for malignant glioma (e.g., single-fraction stereotaxic radiotherapy or brachytherapy)

  * Prior stereotactic radiosurgery boost as part of the initial fractionated external beam radiotherapy regimen allowed

Surgery

* See Disease Characteristics

Other

* Recovered from prior therapy
* No prior investigational intracerebral agents
* At least 4 weeks since prior systemic investigational agents
* No prior localized antitumor therapy for malignant glioma
* No concurrent anticoagulants or antiplatelet therapy, including, but not limited to, any of the following:

  * Heparin
  * Fractionated heparin
  * Warfarin
  * Aspirin
  * Ticlopidine
  * Clopidogrel
  * Dipyridamole
* No other concurrent investigational agents

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2005-10

PRIMARY OUTCOMES:
Toxicities from the start of infusion through the dose limiting toxicity observation period(Phase I) | Start of IL13-PE38QQR infusion to Day 35 or Day 75
  Toxicities reported are those occurring from the start of the IL13 infusion after catheter placement to Day 35 (30 days after the end of the infusion) if there are no or mild MRI changes on Day 35 around the catheter tract or tip. If the MRI change on Day 35 indicates moderate or extensive changes around the catheter tract or tip then the toxicities reported are those occurring from the start of the IL13 infusion to Day 75 (70 days after the end of the infusion).
Maximum safe flow rate (Phase I) | Start of IL13-PE38QQR infusion to Day 35 or Day 70
  Two total flow rates of IL13-PE38QQR, 500 uL/hr and 750 uL/hr, will be studied based on a traditional phase I design. Dose-limiting toxicities occurring during the dose-finding period will determine the maximum safe flow rate. The dose-finding period is the start of the IL13 infusion after catheter placement to Day 35 if there are none or mild MRI changes around the catheter tract or tip on Day 35. If there are moderate or extensive MRI changes around the catheter tract or tip on Day 35 then the dose-finding period is from the start of the IL13 infusion to Day 75.
Maximum tolerated infusion concentration (Phase I) | Start of IL13-PE38QQR infusion to Day 35 or Day 70
  Two infusion concentrations of IL13-PE38QQR, .25 ug/mL and .50 ug/mL, will be studied based on a traditional phase I design. Dose-limiting toxicities occurring during the dose-finding period will determine the maximum tolerated infusion concentration. The dose-finding period is the start of the IL13 infusion after catheter placement to Day 35 if there are none or mild MRI changes around the catheter tract or tip on Day 35. If there are moderate or extensive MRI changes around the catheter tract or tip on Day 35 then the dose-finding period is from the start of the IL13 infusion to Day 75.
Survival post initial recurrence or progression at the maximum safe total flow rate and maximum tolerated infusion concentration (Phase II) | Initial progression to date of death from any cause

SECONDARY OUTCOMES:
Progression-free survival (Phase II) | Initial progression to second progression
IL13receptor α2 chain expression status and distribution | Pre-treatment
  Expression of the IL13 receptor α2 chain will be determined by immunohistochemistry analysis of previously banked fixed primary tumor sections in addition to samples obtained during the on-study resection. Expression of the IL13 receptor α2 chain will also be determined by western blot analysis of previously banked fresh frozen primary tumor samples in addition to samples of relapsed fresh frozen tumor obtained during the on-study resection.
Overall safety | Start of IL13-PE38QQR infusion to disease progression or alternative treatment
  Adverse events reported are those occurring from the start of the IL13 infusion after catheter placement to the maximum of disease progression, start of alternative therapy, withdrawal from the study, death, or completion of the follow-up period. Adverse events will be tabulated by first occurrence of the event, by body system, by maximum severity, and by the highest degree of relationship to the study medication.
Tolerability | Start of IL13-PE38QQR infusion to disease progression or alternative treatment
  Adverse events reported are those occurring from the start of the IL13 infusion after catheter placement to the maximum of disease progression, start of alternative therapy, withdrawal from the study, death, or completion of the follow-up period. Adverse events will be tabulated by first occurrence of the event, by body system, by maximum severity, and by the highest degree of relationship to the study medication.

CONTACTS AND LOCATIONS:
Overall Officials: Anuradha Banerjee, MD, Study Chair — University of California, San Francisco